CLINICAL TRIAL: NCT06255548
Title: The Effect of Immersive Virtual Reality and Music on Anxiety, Fear, and Pain During Circumcision Surgery in Children: A Randomized Controlled Trial
Brief Title: Immersive Virtual Reality and Music During Circumcision in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Hamide Nur Çevik Özdemir, Asst.prof., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Afyonkarahisar
Record Dates: First submitted 2024-02-01; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Fear; Anxiety; Child
Keywords: Immersive Virtual Reality; Music; Pain; Circumcision
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled experimental study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor) Triple-blind (i.e., triple-masking) studies are randomized experiments in which the treatment or intervention is unknown to (a) the research participant, (b) the individual(s) who administer the treatment or intervention, and (c) the individual(s) who assess the outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immersive virtual reality group (Experimental): During the circumcision operation, the IVR group received both routine care and VR game. The children were allowed to play the virtual reality game of their choice. The children in the IVR group had an interactive gaming experience for 10 minutes with the game of their choice, using the remote controls while lying on their backs on the operating table during circumcision.
  Interventions: Other: Immersive virtual reality group
- Music group (Experimental): The researcher explained the use of music headphones to the children in the music group. Each child in the music group was allowed to choose the music he wanted to listen to during the circumcision. In the interview with the children in the music group, the type of music they listened to in their daily lives was asked and the music they wanted to listen to during circumcision was determined.
  Interventions: Other: Music group
- Control group (No Intervention): Children in the control group received routine care and no intervention was performed.

INTERVENTIONS:
Other: Immersive virtual reality group — The children in the IVR group were offered two video games from the Oculus Quest gallery. These games were Ocean Rift and Epic Roller Coaster-T-Rex Kingdom. Ocean Rift is the world's first VR water safari park. It has 12 different marine animals such as dolphins, sharks, and turtles and a habitat. Here one can visit a vibrant underwater world that extends all the way to the Arctic and Atlantis. Epic Roller Coaster-T-Rex Kingdom takes one on a roller coaster ride through the Age of Dinosaurs. There are more than 10 species of dinosaurs such as terrestrial, flying, herbivorous and carnivorous.
  Arms: Immersive virtual reality group
Other: Music group — In musical interventions, it is recommended to play music chosen by individuals. Disposable ear pads were used for each child and the headphones were cleaned after each intervention.
  Arms: Music group

SUMMARY:
The goal of this randomized controlled trial is to examine the effectiveness of immersive virtual reality (IVR) and music on children's anxiety, fear, and pain levels during circumcision surgery.

The main question[s] it aims to answer are:

1. Are immersive virtual reality and music interventions effective in reducing children's anxiety and fear levels during circumcision surgery?
2. Are immersive virtual reality and music interventions effective in reducing children's pain levels during circumcision surgery? There were three groups in the study: control group (n:24), immersive virtual reality group (n:24), and music group (n:24). The control group did not undergo any intervention and only the routine procedure of the clinic was performed. The participants in the immersive virtual reality group played an interactive video game. The participants in the music group listened to music of their preference.

DETAILED DESCRIPTION:
Aim: Circumcision is one of the surgical procedures causing fear and pain in children. This study aimed to examine the effectiveness of immersive virtual reality (IVR) and music on children's anxiety, fear, and pain levels during circumcision surgery.

Methods:The participants were divided into three groups: Immersive virtual reality group (n=24), music group (n=24), and control group (n=24). Data were collected using a Participant Information Form, the Children's Anxiety Meter-Scale (CAM-S), the Children's Fear Scale (CFS), and the Wong-Baker Faces Pain Rating Scale (WBS). Anxiety and fear levels of the children were measured before, during, and after the circumcision operation and their pain levels were measured during and after circumcision. The study was conducted in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Descriptive statistics, analysis of variance, t-test, and Duncan and Bonferroni tests were performed for data analysis.

Intervention protocols: As a routine procedure in the clinic where the study was conducted, the children to be circumcised were admitted to the clinic in the morning on the day of the procedure, and routine preparations for the operation were completed. When the children and their families came to the clinic immediately after hospitalization, they were informed about the study by one of the researchers, and their written and verbal consent was obtained. Then the data were collected using an introductory information form, the Children's Anxiety Meter-Scale (CAM-S), and the Children's Fear Scale (CFS). Children who met the selection criteria were divided into groups by randomization method.

After the children in the experimental groups were taken to the waiting room in the operating room, they were informed by the researcher who would perform the intervention. The researcher explained the use of virtual reality glasses to the children in the IVR group and the use of music headphones to the children in the music group. Each child in the music group was allowed to choose the music he wanted to listen to during the circumcision. The children were also informed that the intervention would be stopped if they experienced motion sickness, eye discomfort, headache, or earache. In the interview with the children in the music group, the type of music they listened to in their daily lives was asked and the music they wanted to listen to during circumcision was determined. Each child in the IVR group was allowed to choose the VR game he wanted to play during the circumcision. Routine procedures were applied for the control group.

Intervention phase:In this study, one group received IVR intervention, and the other group received music intervention to distract the child during the circumcision operation. One of the researchers (an academic with a PhD degree in pediatric nursing) was certified as a music therapy practitioner and had knowledge and experience in virtual reality. The interventions were carried out by this researcher. The researcher complied with the principles of medical and surgical asepsis in the operating room. Just before the intervention, the researcher put the virtual reality glasses on the children in the IVR group and gave the remote controls to their hands. The children in the music group wore music headphones.

Circumcision operations were performed in the same operating room setting by the same pediatric surgeon and operating room team (assistant physician, anesthesia technician, three nurses, and the researcher). The thermocautery assisted guillotine technique was performed in all children during circumcision. Each circumcision operation took an average of 15 minutes for all children in the experimental and control groups. This period included the child's entry and exit to and from the operating room. During this period, the parents of all children waited in the waiting room outside the operating room.

During the circumcision operation, the IVR group received both routine care and VR game. The children were allowed to play the virtual reality game of their choice. The children in the IVR group had an interactive gaming experience for 10 minutes with the game of their choice, using the remote controls while lying on their backs on the operating table during circumcision.

The children in the IVR group were offered two video games from the Oculus Quest gallery. These games were Ocean Rift and Epic Roller Coaster-T-Rex Kingdom. Ocean Rift is the world's first VR water safari park. It has 12 different marine animals such as dolphins, sharks, and turtles and a habitat. Here one can visit a vibrant underwater world that extends all the way to the Arctic and Atlantis. Epic Roller Coaster-T-Rex Kingdom takes one on a roller coaster ride through the Age of Dinosaurs. There are more than 10 species of dinosaurs such as terrestrial, flying, herbivorous and carnivorous. The aforementioned VR video games are commercially available and were obtained from the Oculus Quest 2 Store (https://www.oculus.com/experiences/quest/).

A disposable silicone pad was placed on the Oculus Quest before each use. To minimize direct contact with the device, the patients wore disposable headgear and a face mask (personal protective equipment) before use. The parts of the device in contact with children's faces were cleaned before each intervention.

The children in the music group listened to music at the same volume (60 dB), with the same type of headphones, and the same iPad. The children listened to the music of their choice for 10 minutes after wearing the headphones. In musical interventions, it is recommended to play music chosen by individuals. Disposable ear pads were used for each child and the headphones were cleaned after each intervention.

Children in the control group received routine care and no intervention was performed. Anxiety, fear, and pain of the children in the experimental and control groups were re-evaluated 10 minutes after circumcision by the children and an external observer using the Children's Anxiety Meter-Scale (CAM-S), the Children's Fear Scale (CFS), and the Wong-Baker Faces Pain Rating Scale (WBS).

ELIGIBILITY:
Inclusion Criteria:

* Circumcision in a pediatric surgery clinic
* Agreeing to participate in the study
* Having no visual and hearing problems, having no history of surgical intervention, and having no chronic pain or mental health problems

Exclusion Criteria:

* Presence of contraindications for the procedure (hypospadias, epispadias, bleeding disorders, anatomical disorders),
* Use of any painkillers 24 hours before the procedure,
* Presence of communication problems.

Ages: 6 Years to 8 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Statistical difference between groups about anxiety scores | During the procedure approximately 10 minutes
  Implementation of interventions aimed at reducing anxiety in experimental groups.
  Children's Anxiety Meter-Scale:This scale is used in clinical settings to assess children's anxiety during invasive procedures. Scores obtained from the scale range from 0 to 10.
Statistical difference between groups about fear scores | During the procedure approximately 10 minutes
  Implementation of interventions aimed at reducing fear in experimental groups. Children's Fear Scale:This scale is used in clinical settings to assess children's fear during invasive procedures.The scale consists of five gender-neutral facial expressions, ranging from neutral on the far left to extremely fearful on the far right. The evaluation of facial expressions ranges between 0-4 points.
Statistical difference between groups about pain scores | During the procedure approximately 10 minutes
  Implementation of interventions aimed at reducing pain in experimental groups. Wong-Baker Faces Pain Rating Scale:This scale was developed by Wong and Baker to evaluate pain in children aged 3-18. Scores on the numerical rating scale range from 0 to 10. The scale shows a series of faces ranging from a smiling face (0=very happy/no pain) to a crying face (10=high pain)

CONTACTS AND LOCATIONS:
Overall Officials: Hamide Nur Çevik Özdemir, PhD, Principal Investigator — Afyonkarahisar Health Science University Health Science Faculty
Locations (1):
- Afyonkarahisar Health Science University Health Science Faculty, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buyuk ET, Odabasoglu E, Uzsen H, Koyun M. The effect of virtual reality on Children's anxiety, fear, and pain levels before circumcision. J Pediatr Urol. 2021 Aug;17(4):567.e1-567.e8. doi: 10.1016/j.jpurol.2021.04.008. Epub 2021 Apr 21. PMID 34006462
- [Background] Suzan OK, Sahin OO, Baran O. Effect of Puppet Show on Children's anxiety and pain levels during the circumcision operation: A randomized controlled trial. J Pediatr Urol. 2020 Aug;16(4):490.e1-490.e8. doi: 10.1016/j.jpurol.2020.06.016. Epub 2020 Jun 20. PMID 32669215
- [Background] Luo W, Chen C, Zhou W, Cao A, Zhu W, Zhou Y, Xu Z, Wang J, Zhu B. Biophilic virtual reality on children's anxiety and pain during circumcision: A randomized controlled study. J Pediatr Urol. 2023 Apr;19(2):201-210. doi: 10.1016/j.jpurol.2022.10.023. Epub 2022 Oct 20. PMID 36336624
- [Background] Yeniay D, Tamdo An L, Yucak Ozdemir A, Ak An LO, Kay R SU. Effects of Videos and Therapeutic Music on Preoperative Anxiety and Postoperative Anxiety and Pain Levels in Boys Who Undergo Circumcision. J Perianesth Nurs. 2023 Dec;38(6):918-924. doi: 10.1016/j.jopan.2023.04.007. Epub 2023 Aug 16. PMID 37589631
- [Background] Gezginci E, Suluhan D, Caliskan MB. Is tablet-based interactive distraction effective on pain and anxiety during circumcision in children? A randomized controlled trial. Turk J Urol. 2021 Nov;47(6):518-525. doi: 10.5152/tud.2021.21228. PMID 35118971